CLINICAL TRIAL: NCT03490370
Title: Proof of Concept ELectro-Stimulation of Muscles to resolVe Insulin Resistance in NASH (The Elvis Study)
Brief Title: Proof of Concept ELectro-Stimulation of Muscles to resolVe Insulin Resistance in NASH
Acronym: ELVIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Tayside (Other Government)
Responsible Party: Principal Investigator, John Dillon, Professor, NHS Tayside
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017GA07
Record Dates: First submitted 2018-03-27; First posted 2018-04-06 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: NASH - Nonalcoholic Steatohepatitis; Insulin Sensitivity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Proof of concept study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electronic Muscle Stimulation Activity (Experimental): Electro-muscular stimulation using NeuroTrac MyoPlus 2/4. All participants taking part will be allocated to the Electronic Muscle Stimulation Activity (EMS) intervention from baseline for the duration of 12 weeks. There will be 6 EMS sessions of 35mins/per session each week.
  Interventions: Device: Electro-muscular stimulation using NeuroTrac MyoPlus 2/4

INTERVENTIONS:
Device: Electro-muscular stimulation using NeuroTrac MyoPlus 2/4 — In this pilot study we aim to determine if change in the muscle metabolism can resolve insulin resistance in NAFLD through muscle stimulation by using electro-stimulation. We hypothesise that 6x35 minute sessions per week over a 12 week time scale would mimic effects of resistance exercise on metabolic parameters associated with NAFLD and hepatic steatosis. All 20 participants will have the electro-stimulation intervention.

SUMMARY:
Non-alcoholic steato-hepatitis (NASH) affects up to 3% of the population and leads to liver cirrhosis, hepatocellular carcinoma (HCC) and death. The only known treatment is weight loss and exercise. Many patients cannot or will not achieve this with conventional means. The pathogenic process of the disease is insulin resistance which can be reversed relatively quickly with intense exercise or electrical stimulation of muscle. Most patients cannot achieve or sustain the level of aerobic exercise required; resistance exercise is more sustainable and similarly effective. The aim of this pilot study is to investigate whether electro-muscle stimulation, designed to emulate resistance exercise, resolves NASH in patients and moves them to a less dangerous metabolic steady state which should be easier to maintain.

DETAILED DESCRIPTION:
This is a pilot study which will determine if muscle stimulation by using electro-stimulation can mimic resistance exercise and improve insulin resistance and hepatitis steatosis. We aim to recruit up to 20 patients into the study, needing a minimum of 12 subjects suitable for per protocol analysis. The participants will self-administer EMS for 8 -12 weeks. An interim analysis of change in insulin resistance at 8 weeks of study will be undertaken in the first 4 patients, if this shows a clear effect the study period will be shortened to 8 weeks.

Patients with biopsy proven NASH will be approached by their clinician at their routine liver outpatient clinic and provided with study information alongside the contact details of study staff. Patients will be given adequate time (over 24 hours) to consider the study and will be asked to contact research staff by email or telephone supplied on the PIS if they then wish to participate in the study or require further information. An appointment will be arranged to attend for study screening convenient to the patient where a full in-depth discussion will take place prior to consent or any study procedures undertaken.

Study participants will then follow the study pathway as shown in the flow chart, (section 3.2) Study Matrix (3.3) and as described in the study assessments schedule (section 6).

Electro Muscle Stimulation (EMS) will commence at baseline visit, which will take place in the Institute of Motion Analysis & Research centre, Ninewells hospital, 6 sessions per week self-administered at home, of up to 35 minutes duration for up to a total of 12 weeks. Participants will self-administer muscle stimulation via the Neurotrac Myoplus 2/4 device. Manufactured by: Verity Medical Ltd, in compliance with the European Union Medical Device Directive MDD93/42/EEC under the supervision of SGS, Notified Body number 0120. CE 0120.

Custom STIM (stimulation) mode settings will be utilised and locked for safety. Each participant's own tolerance for the settings within regulated parameters will be used to ensure patient comfort but also allow for optimum muscle activity. 4 channels on the device will be used with 2 sets of skin electrodes attached to the medial and lateral aspects of the quadriceps muscles of each leg.

Assessments of Insulin Sensitivity. This will be based around frequently sampled oral Glucose Tolerance test (fsOGTT) which will be performed in the Clinical Research Centre at baseline, week 4, 8 and 12. The fsOGTT will use the 2 hour, seven sample method following glucose administration (22).

Samples will be analysed for glucose, insulin, c-peptide and non-esterified fatty acids (NEFA), using the model described in Man et al (22). For the days leading up to the test patients should eat a normal diet without restriction, fast overnight from 10pm (at least 8 hours), water is allowed. Regular medication may be taken, If any need to be taken with food it may be best to take them after the test. Patients are asked to refrain from smoking, chewing gum or wearing nicotine patches, during the fasting period until after the test is completed. The procedure will last for 2-2½ hours. On the morning of the test patients will be asked to sit comfortably. A peripheral venous cannula will be inserted into a vein in the hand or arm to allow blood samples to be taken before the glucose drink and at 10, 20, 30, 60, 90, 120 minutes afterwards. The glucose drink should be drunk over a maximum of 5 minutes.

Water is allowed after the glucose drink if the patient is thirsty. After the blood tests are complete the cannula will be removed. They will be offered a drink and something to eat at the end of the test and the patient is free to leave.

Assessments of liver steatosis by MRI liver.

The MRI scanning will take place at the Radiology department, Ninewells hospital. The protocol will consist of three sub-sections, namely (i) cardiac MR for studying heart structure and function (30 minutes scanning); (ii) abdominal MR for measuring liver lipid and iron concentrations, and visceral/sub-cutaneous adipose tissue volumes (20 minutes scanning); and (iii) MR elastography for measuring liver fibrosis (30 minutes scanning). For the baseline visit, patient volunteers will undergo (i) and (ii), and for the follow-up visit patient volunteers will undergo (ii) and (iii). This will ensure that the abdominal MR sub-section of the protocol is acquired at both time-points, with a total scan time that will not exceed 50 minutes for any given session.

ELIGIBILITY:
Inclusion Criteria:

* Male/ Female aged 18 - 75
* Able to give informed consent
* Biopsy proven NASH with a NAS (NAFLD activity score) activity score equal to or greater than 3
* A single hepatic diagnosis.

Exclusion Criteria:

* Presence of other causes of Chronic Liver Disease
* Currently or previously decompensated liver disease (ascites, encephalopathy or variceal bleeding)
* Hepatocellular carcinoma (current or previous)
* Malignancy - of any sort except basal cell carcinoma
* Unstable co morbid disease
* Known HIV positive
* Limb amputation
* Implanted electrical device
* Pregnancy, breastfeeding or undertaking fertility treatment
* Type 1 Diabetes Mellitus (Type 2 diabetes mellitus, diet and metformin acceptable for inclusion)
* Alcohol intake above 14 units a week
* Unable to give informed consent
* Unable to attend required study visits.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2020-02-06 (Actual)

PRIMARY OUTCOMES:
Can electro-stimulated muscle activity demonstrate improvement in insulin resistance. | 10 months
  Change from baseline of frequent sampled Oral Glucose Tolerance Testing (fsOGTT) to end of treatment

SECONDARY OUTCOMES:
Can electro-stimulated muscle activity demonstrate improvement in hepatic steatosis | 10 months
  Change from baseline of liver steatosis to end of treatment via Magnetic Resonance

CONTACTS AND LOCATIONS:
Overall Officials: John Dillon, MD, Principal Investigator — NHS Tayside
Locations (1):
- NHS Tayside, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: No